CLINICAL TRIAL: NCT02908685
Title: A Two Part Seamless, Multi-Center Randomized, Placebo-Controlled, Double-Blind Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of Risdiplam (RO7034067) in Type 2 and 3 Spinal Muscular Atrophy Patients
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of Risdiplam (RO7034067) in Type 2 and 3 Spinal Muscular Atrophy (SMA) Participants
Acronym: SUNFISH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: BP39055; 2016-000750-35 (EudraCT Number)
Expanded Access: NCT04256265 (Approved for marketing)
Record Dates: First submitted 2016-09-19; First posted 2016-09-21 (Estimated); Results first posted 2021-06-15 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-03

CONDITIONS: Muscular Atrophy, Spinal
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Risdiplam

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Part 1 Group A: Adolescents and Adults (Risdiplam) (Experimental): Adolescent and adult participants aged 12-25 years will receive risdiplam for at least 12 weeks. Once the placebo-controlled period is completed and Part 2 dose is selected, participants will be switched to Part 2 dose and will be treated in an open-label phase.
  Interventions: Drug: Risdiplam
- Part 1 Group A: Adolescents and Adults (Placebo) (Placebo Comparator): Adolescent and adult participants aged 12-25 years will receive placebo matching to risdiplam for at least 12 weeks. Once placebo-controlled period is completed, participants will be first switched to their cohort risdiplam dose. After the Part 2 dose is selected, participants will be switched to Part 2 dose and will be treated in an open-label phase.
  Interventions: Drug: Placebo; Drug: Risdiplam
- Part 1 Group B: Children (Placebo) (Placebo Comparator): Children aged 2-11 years will receive placebo matching to risdiplam for at least 12 weeks. Once placebo-controlled period is completed, participants will be first switched to their cohort risdiplam dose. After the Part 2 dose is selected, participants will be switched to Part 2 dose and will be treated in an open-label phase.
  Interventions: Drug: Placebo; Drug: Risdiplam
- Part 1 Group B: Children (Risdiplam) (Experimental): Children aged 2-11 years will receive risdiplam for at least 12 weeks. Once the placebo-controlled period is completed and Part 2 dose is selected, participants will be switched to Part 2 dose and will be treated in an open-label phase.
  Interventions: Drug: Risdiplam
- Part 2: Placebo (Placebo Comparator): Participants aged 2-25 years will receive placebo matching to risdiplam for 12 months. After 12 months of treatment with placebo, participants will be switched to risdiplam (5 mg once daily for participants with a body weight (BW) >/=20kg or 0.25 mg/kg for participants with a BW <20) in a blinded manner and participants will continue with treatment until Month 24. After Month 24, participants will be offered the opportunity to enter the open-label phase.
  Interventions: Drug: Placebo; Drug: Risdiplam
- Part 2: Risdiplam (Experimental): Participants aged 2-25 years will receive risdiplam at the dose selected based on the results from Part 1 of the study (5 mg once daily for participants with a body weight (BW) >/=20kg or 0.25 mg/kg for participants with a BW <20 kg), for 24 months. After 24-month treatment, participants will be offered the opportunity to enter the open-label phase.
  Interventions: Drug: Risdiplam

INTERVENTIONS:
Drug: Placebo — Placebo will be administered orally (via mouth) or through a feeding tube (naso-gastric or gastrostomy tube).
  Arms: Part 1 Group A: Adolescents and Adults (Placebo); Part 1 Group B: Children (Placebo); Part 2: Placebo
Drug: Risdiplam — Risdiplam will be administered orally (via mouth) or through a feeding tube (naso-gastric or gastrostomy tube).
  Other Names: RO7034067

SUMMARY:
Multi-center, randomized, double-blind, placebo-controlled study to assess the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy of Risdiplam in adult and pediatric participants with Type 2 and Type 3 SMA. The study consists of two parts, an exploratory dose finding part (Part 1) of Risdiplam for 12 weeks and a confirmatory part (Part 2) of Risdiplam for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of 5q-autosomal recessive SMA
* Negative blood pregnancy test at screening and agreement to comply with measures to prevent pregnancy and restrictions on sperm donation
* For Part 1: Type 2 or 3 SMA ambulant or non-ambulant
* For Part 2: 1) Type 2 or 3 SMA non-ambulant; 2) RULM entry item A greater than or equal to 2; 3) ability to sit independently as assessed by item 9 of the MFM

Exclusion Criteria:

* Concomitant or previous participation in any investigational drug or device study within 90 days prior to screening, or 5 half-lives of the drug, whichever is longer
* Concomitant or previous administration of a SMN2-targeting antisense oligonucleotide, SMN2 splicing modifier or gene therapy either in a clinical study or as part of medical care
* Any history of cell therapy
* Hospitalization for a pulmonary event within the last 2 months or planned at time of screening
* Surgery for scoliosis or hip fixation in the one year preceding screening or planned within the next 18 months
* Unstable gastrointestinal, renal, hepatic, endocrine, or cardiovascular system diseases as considered to be clinically significant by the Investigator
* Presence of clinically significant electrocardiogram abnormalities before study drug administration from average of triplicate measurement or cardiovascular disease indicating a safety risk for participants as determined by the Investigator
* Any major illness within one month before the screening examination or any febrile illness within one week prior to screening and up to first dose administration
* Recently initiated treatment (within less than [<] 6 months prior to randomization) with oral salbutamol or another beta 2-adrenergic agonist taken orally
* Any prior use of chloroquine, hydroxychloroquine, retigabin, vigabatrin or thioridazine, is not allowed
* Ascertained or presumptive hypersensitivity (e.g., anaphylactic reaction) to Risdiplam or to the constituents of its formulation
* Recent history (less than one year) of ophthalmological diseases
* Participants requiring invasive ventilation or tracheostomy

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 231 (Actual)
Dates: Start 2016-10-19 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2023-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (45):
- United States (2):
  - Stanford University Medical Center, Palo Alto, California
  - Columbia University Medical Center; The Neurological Institute of New York, New York, New York
- Belgium (3):
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
  - Chr de La Citadelle, Liège
- Instituto de Puericultura E Pediatria Martagão Gesteira, Rio de Janeiro, Rio de Janeiro, Brazil
- Canada (3):
  - Alberta Children's Hospital Division of Pediatric Neurology, Calgary, Alberta
  - London Health Sciences Centre; Children's Hospital; Pediatrics, London, Ontario
  - McGill University Health Centre - Glen Site, Montreal, Quebec
- China (2):
  - Peking University First Hospital, Beijing
  - Children's Hospital of Fudan University, Shanghai
- Clinical Medical Center Zagreb; University Hospital Rebro Department of Paediatrics, Zagreb, Croatia
- France (5):
  - Hopital Femme Mere Enfant; Medecine Physique et Readaptation Pediatrique ? L?ESCALE, Bron
  - Hopital Roger Salengro, Lille
  - CHU de Nantes - Hotel Dieu, Nantes
  - Hôpital Necker-Enfants Malades; Service de neuropédiatrie, Paris
  - Hopital Armand Trousseau, Paris
- Universitätsklinikum Freiburg; Klinik für Neuropädiatrie und Muskelerkrankungen, Freiburg im Breisgau, Germany
- Italy (5):
  - IRCCS Ospedale Pediatrico Bambino Gesù; U.O. Malattie Neuromuscolari e Neurodegenerative, Rome, Lazio
  - Policlinico Agostino Gemelli; Dipartimento di Neuropsichiatria Infantile, Rome, Lazio
  - IRCCS Istituto Giannina Gaslini; U.O.S.D. Centro di Miologia e Patologie Neurodegenerative, Genoa, Liguria
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico; Unità Operativa Complessa di Neurologia, Milan, Lombardy
  - Fondazione IRCCS Istituto Neurologico ?Carlo Besta?; UO di Neurologia dello Sviluppo, Milan, Lombardy
- Japan (10):
  - Fukuoka Children's Hospital, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - Hyogo Medical University Hospital, Hyōgo
  - Minami Kyushu National Hospital, Kagoshima
  - Miyagi Children's Hospital, Miyagi
  - Shiga Medical Center for Children, Shiga
  - Shizuoka Children's Hospital, Shizuoka
  - Jichi Medical University Hospital, Tochigi
  - Center Hospital of the National Center for Global Health and Medicine, Tokyo
  - National Center Of Neurology And Psychiatry Hospital, Tokyo
- Poland (3):
  - Szpital Gdanskiego Uniwersytetu Medycznego; Clinic of developmental neurology, Gda?sk
  - Uniwersytecki Szpital Kliniczny w Poznaniu; Od. Kliniczny Neurologii Dzieci i M?odziezy, Późna
  - Klinika Neurologii I Wydzialu Lekarskiego WUM w Warszawie, Warsaw
- Russian Children Neuromuscular Center of Veltischev, Moscow, Moscow Oblast, Russia
- Clinic for Neurology and Psychiatry for Children and Youth, Belgrade, Serbia
- Spain (4):
  - Hospital Sant Joan De Deu, Esplugues de Llobregas, Barcelona
  - Hospital Universitari Vall d'Hebron; Servicio de Reumatologia, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
- Turkey (Türkiye) (2):
  - Hacettepe University, School of Medicine; Pediatrics Department; Pediatrics Child Neurology Unit, Ankara
  - Hospital Yeditepe University Kozyatagi; Pediatry, Atasehir- Istanbul
- University of Oxford; Department of Paediatrics, Headington, United Kingdom

REFERENCES:
- [Derived] Cleary Y, Kletzl H, Grimsey P, Heinig K, Ogungbenro K, Silber Baumann HE, Frey N, Aarons L, Galetin A, Gertz M. Estimation of FMO3 Ontogeny by Mechanistic Population Pharmacokinetic Modelling of Risdiplam and Its Impact on Drug-Drug Interactions in Children. Clin Pharmacokinet. 2023 Jun;62(6):891-904. doi: 10.1007/s40262-023-01241-7. Epub 2023 May 6. PMID 37148485
- [Derived] Mercuri E, Deconinck N, Mazzone ES, Nascimento A, Oskoui M, Saito K, Vuillerot C, Baranello G, Boespflug-Tanguy O, Goemans N, Kirschner J, Kostera-Pruszczyk A, Servais L, Gerber M, Gorni K, Khwaja O, Kletzl H, Scalco RS, Staunton H, Yeung WY, Martin C, Fontoura P, Day JW; SUNFISH Study Group. Safety and efficacy of once-daily risdiplam in type 2 and non-ambulant type 3 spinal muscular atrophy (SUNFISH part 2): a phase 3, double-blind, randomised, placebo-controlled trial. Lancet Neurol. 2022 Jan;21(1):42-52. doi: 10.1016/S1474-4422(21)00367-7. PMID 34942136
- See also: roche-sma-clinicaltrials.com provides information about the Roche Sunfish clinical trial NCT02908685 and molecule being investigated in SMA. — http://roche-sma-clinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Part 1 was conducted at 5 investigational sites across 4 countries, and Part 2 was conducted at 42 investigational sites across 14 countries. Screening in both Part 1 and 2 was up to 30 days prior to first dose.
Pre-assignment Details: In Part 1 participants were initially enrolled by age and in a dose-escalating design; each group included participants on active and placebo treatment in a 2:1 ratio. After Part 2 dose selection the study enrolled additional participants in a 2:1 ratio in Part 2.
Groups:
- Part 1 Group A Cohort 1: Adolescents and Adults (3 mg Risdiplam); Part 1 Group A Cohort 2: Adolescents and Adults (5 mg Risdiplam): Adolescent and adult participants aged 12-25 years received risdiplam for at least 12 weeks. Once the placebo-controlled period was completed and Part 2 dose was selected, participants switched to Part 2 dose and were treated in an open-label phase.
- Part 1 Group A Cohort 1: Adolescents and Adults (Placebo): Adolescent and adult participants aged 12-25 years received placebo matching to risdiplam for at least 12 weeks. Once the placebo-controlled period was completed, participants first switched to their cohort risdiplam dose (i.e. 3 mg). After the Part 2 dose was selected, participants switched to Part 2 dose and were treated in an open-label phase.
- Part 1 Group A Cohort 2: Adolescents and Adults (Placebo): Adolescent and adult participants aged 12-25 years received placebo matching to risdiplam for at least 12 weeks. Once the placebo-controlled period was completed, participants first switched to their cohort risdiplam dose (i.e. 5 mg). After the Part 2 dose was selected, participants switched to Part 2 dose and were treated in an open-label phase.
- Part 1 Group B Cohort 1: Children (0.02 mg/kg Risdiplam): Children aged 2-11 years received risdiplam for at least 12 weeks. During the placebo-controlled period, participants escalated to 0.05 mg/kg and then to 0.15 mg/kg in two steps. Once the placebo-controlled period was completed, and after Part 2 dose was selected, participants switched to Part 2 dose and were treated in an open-label phase.
- Part 1 Group B Cohort 2: Children (0.05 mg/kg Risdiplam): Children aged 2-11 years received risdiplam for at least 12 weeks. During the placebo-controlled period, participants escalated to 0.15 mg/kg in one step. Once the placebo-controlled period was completed, and after Part 2 dose was selected, participants switched to Part 2 dose and were treated in an open-label phase.
- Part 1 Group B Cohort 3: Children (0.25 mg/kg Risdiplam): Children aged 2-11 years received risdiplam for at least 12 weeks. Once the placebo-controlled period was completed, and after Part 2 dose was selected, participants switched to Part 2 dose and were treated in an open-label phase.
- Part 1 Group B Cohort 1: Children (Placebo); Part 1 Group B Cohort 2: Children (Placebo): Children aged 2-11 years received placebo matching to risdiplam for at least 12 weeks. Once the placebo-controlled period was completed, participants first switched to the final 0.15 mg/kg cohort risdiplam dose. After the Part 2 dose was selected, participants switched to Part 2 dose and were treated in an open-label phase.
- Part 1 Group B Cohort 3: Children (Placebo): Children aged 2-11 years received placebo matching to risdiplam for at least 12 weeks. Once the placebo-controlled period was completed, and after Part 2 dose was selected, participants switched to Part 2 dose and were treated in an open-label phase.
- Part 1 Group A: OLE: Once the placebo-controlled period was completed and Part 2 dose was selected, adolescents and adults switched to Part 2 dose and were treated in an open-label extension (OLE) phase.
- Part 1 Group B: OLE: Once the placebo-controlled period was completed and Part 2 dose was selected, children switched to Part 2 dose and were treated in an open-label extension (OLE) phase.
- Part 2: Risdiplam: Participants aged 2-25 years received risdiplam at the dose of 5 mg once daily for participants with a body weight (BW) >/=20kg or 0.25 mg/kg for participants with a BW <20 kg for 12 months. Once the Part 2 placebo-controlled period was completed participants received risdiplam at the same dose level for another 12 months (Month 12-24) in the open-label treatment (OLT) phase. After Month 24 participants entered the Part 2 OLE phase and continued to receive risdiplam at the same dose level.
- Part 2: Placebo: Participants aged 2-25 years received placebo matching to risdiplam for 12 months. After 12 months of treatment with placebo, participants switched to risdiplam (5 mg once daily for participants with a body weight (BW) >/=20kg or 0.25 mg/kg for participants with a BW <20) in a blinded manner in the OLT phase. After Month 24 participants entered the Part 2 OLE phase and continued to receive risdiplam at the same dose level.
Period: Part 1 Placebo-Controlled
Arm/Group | Part 1 Group A Cohort 1: Adolescents and Adults (3 mg Risdiplam) | Part 1 Group A Cohort 2: Adolescents and Adults (5 mg Risdiplam) | Part 1 Group A Cohort 1: Adolescents and Adults (Placebo) | Part 1 Group A Cohort 2: Adolescents and Adults (Placebo) | Part 1 Group B Cohort 1: Children (0.02 mg/kg Risdiplam) | Part 1 Group B Cohort 2: Children (0.05 mg/kg Risdiplam) | Part 1 Group B Cohort 3: Children (0.25 mg/kg Risdiplam) | Part 1 Group B Cohort 1: Children (Placebo) | Part 1 Group B Cohort 2: Children (Placebo) | Part 1 Group B Cohort 3: Children (Placebo) | Part 1 Group A: OLE | Part 1 Group B: OLE | Part 2: Risdiplam | Part 2: Placebo
Started | 7 | 7 | 3 | 3 | 7 | 7 | 7 | 3 | 4 | 3 | 0 | 0 | 0 | 0
Completed | 7 | 7 | 3 | 3 | 7 | 7 | 7 | 3 | 4 | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1 OLE
Arm/Group | Part 1 Group A Cohort 1: Adolescents and Adults (3 mg Risdiplam) | Part 1 Group A Cohort 2: Adolescents and Adults (5 mg Risdiplam) | Part 1 Group A Cohort 1: Adolescents and Adults (Placebo) | Part 1 Group A Cohort 2: Adolescents and Adults (Placebo) | Part 1 Group B Cohort 1: Children (0.02 mg/kg Risdiplam) | Part 1 Group B Cohort 2: Children (0.05 mg/kg Risdiplam) | Part 1 Group B Cohort 3: Children (0.25 mg/kg Risdiplam) | Part 1 Group B Cohort 1: Children (Placebo) | Part 1 Group B Cohort 2: Children (Placebo) | Part 1 Group B Cohort 3: Children (Placebo) | Part 1 Group A: OLE | Part 1 Group B: OLE | Part 2: Risdiplam | Part 2: Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 31 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 30 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Period: Part 2 Placebo-Controlled: Month 1-12
Arm/Group | Part 1 Group A Cohort 1: Adolescents and Adults (3 mg Risdiplam) | Part 1 Group A Cohort 2: Adolescents and Adults (5 mg Risdiplam) | Part 1 Group A Cohort 1: Adolescents and Adults (Placebo) | Part 1 Group A Cohort 2: Adolescents and Adults (Placebo) | Part 1 Group B Cohort 1: Children (0.02 mg/kg Risdiplam) | Part 1 Group B Cohort 2: Children (0.05 mg/kg Risdiplam) | Part 1 Group B Cohort 3: Children (0.25 mg/kg Risdiplam) | Part 1 Group B Cohort 1: Children (Placebo) | Part 1 Group B Cohort 2: Children (Placebo) | Part 1 Group B Cohort 3: Children (Placebo) | Part 1 Group A: OLE | Part 1 Group B: OLE | Part 2: Risdiplam | Part 2: Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 120 | 60
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 117 | 59
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Not completed — Changed to Spinraza | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Changed to other treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Part 2 OLT: Month 12-24
Arm/Group | Part 1 Group A Cohort 1: Adolescents and Adults (3 mg Risdiplam) | Part 1 Group A Cohort 2: Adolescents and Adults (5 mg Risdiplam) | Part 1 Group A Cohort 1: Adolescents and Adults (Placebo) | Part 1 Group A Cohort 2: Adolescents and Adults (Placebo) | Part 1 Group B Cohort 1: Children (0.02 mg/kg Risdiplam) | Part 1 Group B Cohort 2: Children (0.05 mg/kg Risdiplam) | Part 1 Group B Cohort 3: Children (0.25 mg/kg Risdiplam) | Part 1 Group B Cohort 1: Children (Placebo) | Part 1 Group B Cohort 2: Children (Placebo) | Part 1 Group B Cohort 3: Children (Placebo) | Part 1 Group A: OLE | Part 1 Group B: OLE | Part 2: Risdiplam | Part 2: Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 117 | 59
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 116 | 59
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Part 2 OLE: > Month 24
Arm/Group | Part 1 Group A Cohort 1: Adolescents and Adults (3 mg Risdiplam) | Part 1 Group A Cohort 2: Adolescents and Adults (5 mg Risdiplam) | Part 1 Group A Cohort 1: Adolescents and Adults (Placebo) | Part 1 Group A Cohort 2: Adolescents and Adults (Placebo) | Part 1 Group B Cohort 1: Children (0.02 mg/kg Risdiplam) | Part 1 Group B Cohort 2: Children (0.05 mg/kg Risdiplam) | Part 1 Group B Cohort 3: Children (0.25 mg/kg Risdiplam) | Part 1 Group B Cohort 1: Children (Placebo) | Part 1 Group B Cohort 2: Children (Placebo) | Part 1 Group B Cohort 3: Children (Placebo) | Part 1 Group A: OLE | Part 1 Group B: OLE | Part 2: Risdiplam | Part 2: Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 116 | 59
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 103 | 53
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 6
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Reason not specified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Part 2: Risdiplam: Participants aged 2-25 years received risdiplam at the dose of 5 mg once daily for participants with a body weight (BW) >/=20kg or 0.25 mg/kg for participants with a BW <20 kg for 12 months.
- Part 2: Placebo: Participants aged 2-25 years received placebo matching to risdiplam for 12 months. After 12 months of treatment with placebo, participants switched to risdiplam (5 mg once daily for participants with a body weight (BW) >/=20kg or 0.25 mg/kg for participants with a BW <20) in a blinded manner and participants will continue with treatment and observations.
- Total: Total of all reporting groups
Arm/Group | Part 1 Group A Cohort 1: Adolescents and Adults (3 mg Risdiplam) | Part 1 Group A Cohort 2: Adolescents and Adults (5 mg Risdiplam) | Part 1 Group A Cohort 1: Adolescents and Adults (Placebo) | Part 1 Group A Cohort 2: Adolescents and Adults (Placebo) | Part 1 Group B Cohort 1: Children (0.02 mg/kg Risdiplam) | Part 1 Group B Cohort 2: Children (0.05 mg/kg Risdiplam) | Part 1 Group B Cohort 3: Children (0.25 mg/kg Risdiplam) | Part 1 Group B Cohort 1: Children (Placebo) | Part 1 Group B Cohort 2: Children (Placebo) | Part 1 Group B Cohort 3: Children (Placebo) | Part 2: Risdiplam | Part 2: Placebo | Total
Number analyzed (Participants) | 7 | 7 | 3 | 3 | 7 | 7 | 7 | 3 | 4 | 3 | 120 | 60 | 231
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Intent-to-Treat (ITT) population: Part 1 and Part 2 were analyzed separately and population results are provided for each part in the study.
  Years
    Part 1: number analyzed (Participants) | 7 | 7 | 3 | 3 | 7 | 7 | 7 | 3 | 4 | 3 | 0 | 0 | 51
    Part 1 | 13.3 (1.1) | 18.1 (4.6) | 14.7 (1.5) | 17.3 (5.1) | 6.1 (2.9) | 4.3 (1.7) | 6.0 (2.7) | 5.3 (2.1) | 3.5 (0.6) | 5.3 (2.9) |  |  | 9.4 (6.0)
    Part 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 120 | 60 | 180
    Part 2 |  |  |  |  |  |  |  |  |  |  | 9.9 (5.8) | 10.3 (6.0) | 10.0 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 1 | 2 | 5 | 3 | 4 | 0 | 2 | 0 | 61 | 30 | 118
  Male | 2 | 2 | 2 | 1 | 2 | 4 | 3 | 3 | 2 | 3 | 59 | 30 | 113
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 23 | 12 | 36
  White | 7 | 7 | 3 | 3 | 6 | 6 | 7 | 3 | 3 | 3 | 80 | 41 | 169
  Multiple | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 3
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 7 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 7
  Not Hispanic or Latino | 7 | 7 | 3 | 3 | 6 | 7 | 7 | 3 | 4 | 3 | 114 | 57 | 221
  Not Stated | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Selected Part 2 Dose of Risdiplam for Participants With a Body Weight (BW) of >/=20kg
Description: The Internal Monitoring Committee (IMC) was responsible for selecting the dose for Part 2 of the study (pivotal dose). An external Independent Data Monitoring Committee (iDMC) reviewed data from Part 1 and confirmed the dose-selection decision of the IMC. The dose for Part 2 selected by the IMC was a dose that: 1.Was judged to be safe and well-tolerated, based on all available safety data from Part 1 and as confirmed by the iDMC; 2. Resulted in an exposure at steady-state below the exposure cap (mean value) of AUC0-24h,ss 2000 ng*h/mL (adjusted for free-fraction, if required); 3. Resulted in an SMN protein increase that was expected to be clinically relevant.
Time Frame: Day 1 up to at least 4 weeks on study (Up to CCOD of 25 July 2017)
Population: All participants in Part 1.
Measure: Number; unit: milligram (mg)
Groups:
- Part 1: All Risdiplam: Children aged 2-11 years and adolescent and adult participants aged 12-25 years received risdiplam or risdiplam matching placebo.
Arm/Group | Part 1: All Risdiplam
Number analyzed (Participants) | 51
milligram (mg) | 5

2. Primary Outcome: Part 1: Selected Part 2 Dose of Risdiplam for Participants With BW of <20kg
Description: as for outcome 1
Time Frame: Day 1 up to at least 4 weeks on study (Up to CCOD of 25 July 2017)
Population: All participants in Part 1.
Measure: Number; unit: milligram/kilogram (mg/kg)
Arm/Group | Part 1: All Risdiplam
Number analyzed (Participants) | 51
milligram/kilogram (mg/kg) | 0.25

3. Primary Outcome: Part 2: Change From Baseline in the Total Motor Function Measure 32 (MFM-32) Total Score at Month 12
Description: The Motor Function Measure 32 (MFM32) is a scale constructed for use in neuromuscular disorders. It comprises 32 items that evaluate physical function in three dimensions: D1 function related to standing and transfer; D2 axial and proximal function; D3 distal motor function. Tasks are scored with a 4-point Likert scale: 0 - cannot initiate the task or maintain the starting position; 1 - performs the task partially; 2 - performs the task incompletely or imperfectly; 3 - performs the task fully and "normally". The 32 scores are summed and expressed on a 0-100 scale for the MFM32 total score. Higher scores indicate increased motor function. A positive change from Baseline indicates improvement. MMRM analysis was performed based on primary efficacy hypothetical estimand, which included participants data assuming no prohibited medication intended for treatment of SMA was received and participants continued on their randomized treatment until the analysis time point at Month 12.
Time Frame: Baseline (Day-1) and Month 12
Population: The intent-to-treat (ITT) population defined as all randomized participants in Part 2. Participants with missing MFM32 total score at Baseline were not included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 115 | 59
Scores on a Scale | 1.36 [0.61 to 2.11] | -0.19 [-1.22 to 0.84]
Statistical Analysis 1: Comparison: Part 2: Risdiplam vs Part 2: Placebo; Test type: Superiority — This is the first end point and first family tested in the hierarchical testing. The variables included in the MMRM model are: baseline total score, treatment, age group, visit, treatment-by-visit and baseline score-by-visit interaction; p = 0.0156, Mixed Model Repeated Measure Analysis; Least Square Mean Difference = 1.55, 95% CI 2-sided [0.30 to 2.81]

4. Secondary Outcome: Part 2: Percentage of Participants With Marked Improvement (Defined as >= 3) in the Total Motor Function Measure (MFM32) Score at Month 12
Description: The MFM32 comprises 32 items that evaluate physical function. The scoring of each task uses a 4-point Likert scale: 0 - cannot initiate the task or maintain the starting position; 1 - performs the task partially; 2 - performs the task incompletely or imperfectly; 3 - performs the task fully and "normally". The 32 scores are summed and expressed on a 0-100 scale for the MFM32 total score. A change in MFM32 total score of threshold >/=3 represents marked improvement in this measure. Logistic regression analysis was performed based on efficacy hypothetical estimand, which included participants data assuming no prohibited medication intended for treatment of SMA was received and participants continued on their randomized treatment until the analysis time point at Month 12.
Time Frame: At Month 12
Population: The intent-to-treat (ITT) population defined as all randomized participants in Part 2. Participants with missing MFM32 total score at Baseline were not included in the analysis. Missing results at Month 12 are considered as non-responders.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 115 | 59
Percentage of Participants | 38.3 [28.94 to 47.58] | 23.7 [12.03 to 35.43]
Statistical Analysis 1: Comparison: Part 2: Risdiplam vs Part 2: Placebo; Test type: Superiority — This is the second end point and second family tested in the hierarchical testing. Logistic Regression Model.The variables included in the logistic regression are: baseline total score, treatment and age group; p = 0.0469, Wald test — Adjusted p-Value The adjusted p-values were derived based on all the p-values from end points in order of the hierarchical testing up to the current endpoint; Odds Ratio (OR) = 2.35, 95% CI 2-sided [1.01 to 5.44]

5. Secondary Outcome: Part 2: Change From Baseline in the Total Score of the Revised Upper Limb Module (RULM) at Month 12
Description: The RULM is a 20 items scale that assesses the proximal and distal motor functions of the arm. There is an entry item and the remaining 18 items are scored on the 3 point scale of: 0: cannot complete task independently; 1: modified method but can complete task independently; 2: completes task without any assistance, and with 1 item scored on a 2 point scale of as a can/cannot score with 1 as the highest score. The RULM total score is the sum of 19 items scores with range of 0-37, and the entry item does not contribute to the total score. Higher scores indicate greater upper limb function. A positive change from Baseline indicates improvement. MMRM analysis was performed based on the efficacy hypothetical estimand, which included participants data assuming no prohibited medication intended for treatment of SMA was received and participants continued on their randomized treatment until the analysis time point at Month 12.
Time Frame: Baseline (Day-1) and Month 12
Population: The intent-to-treat (ITT) population defined as all randomized participants in Part 2. Participants with missing RULM total score at Baseline were not included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 119 | 58
Scores on a Scale | 1.61 [1.00 to 2.22] | 0.02 [-0.83 to 0.87]
Statistical Analysis 1: Comparison: Part 2: Risdiplam vs Part 2: Placebo; Test type: Superiority — This is the third end point and third family tested in the hierarchical testing. The variables included in the MMRM model are: baseline total score, treatment, age group, visit, treatment-by-visit and baseline score-by-visit interaction; p = 0.0469, Mixed Model Repeated Measure Analysis — [p-value comment as in outcome 4, analysis 1]; Least Square Mean Difference = 1.59, 95% CI 2-sided [0.55 to 2.62]

6. Secondary Outcome: Part 2: Change From Baseline in Total Score of Hammersmith Functional Motor Scale Expanded (HFMSE) at Month 12
Description: The HFMSE scale contains 33 items, which are scored on a 3-point Likert-type scale (0-2) and summed to derive the total score, with lower scores indicating greater impairment. The HFMSE contains a series of assessments designed to assess important functional abilities, including standing, transfers, ambulation, and proximal and axial function. The overall score is the sum of the scores for all activities with a maximum achievable score of 66. Higher scores indicate greater motor function. A positive change from Baseline indicates improvement. MMRM analysis was performed based on the efficacy hypothetical estimand, which included participants data assuming no prohibited medication intended for treatment of SMA was received and participants continued on their randomized treatment until the analysis time point at Month 12.
Time Frame: Baseline (Day-1) and Month 12
Population: The intent-to-treat (ITT) population defined as all randomized participants in Part 2.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 120 | 60
Scores on a Scale | 0.95 [0.29 to 1.61] | 0.37 [-0.54 to 1.28]
Statistical Analysis 1: Comparison: Part 2: Risdiplam vs Part 2: Placebo; Test type: Superiority — This is one of the two end points in family four in the hierarchical testing. The variables included in the MMRM model are: baseline total score, treatment, age group, visit, treatment-by-visit and baseline score-by-visit interaction; p = 0.3902, Mixed Model Repeated Measure Analysis — [p-value comment as in outcome 4, analysis 1]; Least Square Mean Difference = 0.58, 95% CI 2-sided [-0.53 to 1.69]

7. Secondary Outcome: Part 2: Change From Baseline in Forced Vital Capacity (FVC) at Month 12 in Participants Aged 6-25 Years
Description: Spirometry is a pulmonary function test that assesses how the lungs work by measuring how much air moves through the airways. Spirometry was performed by all participants aged 6 or older. Forced vital capacity (FVC) is the total volume that can be exhaled after inhaling maximally. The best % predicted value out of all attempts were used for the analysis. MMRM analysis was performed based on the efficacy hypothetical estimand, which included participants data assuming no prohibited medication intended for treatment of SMA was received and participants continued on their randomized treatment until the analysis time point at Month 12.
Time Frame: Baseline (Day-1) and Month 12
Population: The intent-to-treat (ITT) population defined as all randomized participants in Part 2. Participants with missing FVC data at Baseline were not included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Predicted
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 83 | 40
Percentage Predicted | -5.16 [-7.93 to -2.39] | -3.11 [-6.59 to 0.74]
Statistical Analysis 1: Comparison: Part 2: Risdiplam vs Part 2: Placebo; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.3902, Mixed Model Repeated Measure Analysis — [p-value comment as in outcome 4, analysis 1]; Least Square Mean Difference = -2.05, 95% CI 2-sided [-6.67 to 2.56]

8. Secondary Outcome: Part 2: Change From Baseline in the Caregiver-Reported SMA Independence Scale (SMAIS) Total Score at Month 12
Description: The SMA Independence Scale (SMAIS) was developed specifically for SMA participants in order to assess function-related independence. The SMAIS contains 29 items, assessing the amount of assistance required from another individual to perform daily activities such as eating, or bathing. Each item is scored on a 0-4 scale (with an additional option to indicate that an item is non-applicable). The SMAIS total score ranging from 0-44 is obtained based on 22 items with each item on the 0-2 scale. Lower scores indicate greater dependence on another individual. The SMAIS was completed by participants aged 12 years or older and caregivers of participants aged 2-25 years. MMRM analysis was performed based on efficacy hypothetical estimand, which included participants data assuming no prohibited medication intended for treatment of SMA was received and participants continued on their randomized treatment until the analysis time point at Month 12.
Time Frame: Baseline (Day-1) and Month 12
Population: The intent-to-treat (ITT) population defined as all randomized participants in Part 2. Participants with missing SMAIS total score at Baseline were not included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 116 | 60
Scores on a Scale | 1.65 [0.66 to 2.63] | -0.91 [-2.23 to 0.42]
Statistical Analysis 1: Comparison: Part 2: Risdiplam vs Part 2: Placebo; Test type: Superiority — This is the sixth endpoint and the fifth family tested in the hierarchical testing. The variables included in the MMRM model are: baseline total score, treatment, age group, visit, treatment-by-visit and baseline score-by-visit interaction; p = 0.3902, Mixed Model Repeated Measure Analysis — [p-value comment as in outcome 4, analysis 1]; Least Square Mean Difference = 2.55, 95% CI 2-sided [0.93 to 4.17]

9. Secondary Outcome: Part 2: Percentage of Participants Rated by Clinicians as Improved in the Clinical Global Impression of Change (CGI-C) Scale Ratings at Month 12
Description: The Clinical Global Impression of Change (CGI-C) is used to score a clinician's impression of a participant's change in global health. The CGI-C is a single item measure of change in global health, using seven response options: "very much improved", "much improved", "minimally improved", "no change", "minimally worse", "much worse", and "very much worse". Participants considered as "improved" included responses of "very much improved, "much improved" and "minimally improved". Logistic regression analysis was performed based on efficacy hypothetical estimand, which included participants data assuming no prohibited medication intended for treatment of SMA was received and participants continued on their randomized treatment until the analysis time point at Month 12.
Time Frame: At Month 12
Population: The intent-to-treat (ITT) population defined as all randomized participants in Part 2. Missing results at Month 12 are considered as non-responders.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 120 | 60
Percentage of Participants | 47.5 [38.15 to 56.86] | 40.0 [26.77 to 53.23]
Statistical Analysis 1: Comparison: Part 2: Risdiplam vs Part 2: Placebo; CGI Improved; Test type: Superiority — This is the seventh endpoint and the sixth family tested in the hierarchical testing. Logistic Regression Model. The variables included in the logistic regression are: baseline total score, treatment and age group; p = 0.3902, Wald-test — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.70 to 2.74]

10. Secondary Outcome: Part 2: Percentage of Participants Who Achieve Stabilization or Improvement (Defined as >= 0) in the Total Motor Function Measure (MFM-32) Score at Month 12
Description: The MFM32 comprises 32 items that evaluate physical function in three dimensions: D1 function related to standing and transfer; D2 axial and proximal function; D3 distal motor function. Tasks are scored with a 4-point Likert scale: 0 - cannot initiate the task or maintain the starting position; 1 - performs the task partially; 2 - performs the task incompletely or imperfectly; 3 - performs the task fully and "normally". The 32 scores are summed and expressed on a 0-100 scale for the MFM32 total score. Higher scores indicate increased motor function. Logistic regression analysis was performed based on efficacy hypothetical estimand, which included participants data assuming no prohibited medication intended for treatment of SMA was received and participants continued on their randomized treatment until the analysis time point at Month 12.
Time Frame: At Month 12
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 115 | 59
Percentage of Participants | 69.6 [60.72 to 78.41] | 54.2 [40.68 to 67.80]
Statistical Analysis 1: Comparison: Part 2: Risdiplam vs Part 2: Placebo; Test type: Superiority — Logistic Regression Model. The variables included in the logistic regression are: baseline total score, treatment and age group; p = 0.0430, Wald test; Odds Ratio (OR) = 2.00, 95% CI 2-sided [1.02 to 3.93]

11. Secondary Outcome: Part 2: Percentage of Participants Who Achieve an Improvement of at Least One Standard Error of Measurement on the Total MFM-32 Score at Month 12
Description: The MFM32 comprises 32 items that evaluate physical function in three dimensions: D1 standing and transfer; D2 axial and proximal function; D3 distal motor function. Tasks are scored with a 4-point Likert scale: 0-cannot initiate the task or maintain the starting position; 1-performs the task partially; 2-performs the task incompletely or imperfectly; 3-performs the task fully and "normally". The 32 scores are summed and expressed on a 0-100 scale for the total score. Higher scores indicate increased motor function. Standard error of measurement (SEM) is derived using 32 items scores and total scores at baseline. Change from baseline > = one SEM is equivalent to a change >= 4. Logistic regression analysis was performed based on efficacy hypothetical estimand included participants data assuming no prohibited medication intended for treatment of SMA was received and participants continued on their randomized treatment until the analysis time point at Month 12.
Time Frame: At Month 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 115 | 59
Percentage of Participants | 28.7 [20.65 to 37.88] | 16.9 [8.44 to 28.97]

12. Secondary Outcome: Part 2: Change From Baseline in the MFM-32 Domain 1 (D1) Score at Month 12
Description: The MFM32 comprises 32 items that evaluate physical function in three dimensions: D1 function related to standing and transfer; D2 axial and proximal function; D3 distal motor function. Tasks are scored with a 4-point Likert scale: 0 - cannot initiate the task or maintain the starting position; 1 - performs the task partially; 2 - performs the task incompletely or imperfectly; 3 - performs the task fully and "normally". The D1 items score are summed and expressed on 0-100 scale for the MFM D1 total score. Higher scores indicate increased motor function. A positive change from Baseline indicates improvement. MMRM analysis was performed based on efficacy hypothetical estimand, which included participants data assuming no prohibited medication intended for treatment of SMA was received and participants continued on their randomized treatment until the analysis time point at Month 12.
Time Frame: Baseline (Day-1) and Month 12
Population: The intent-to-treat (ITT) population defined as all randomized participants in Part 2. Participants with missing MFM32 D1 score at Baseline were not included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 118 | 60
Scores on a Scale | 0.37 [-0.12 to 0.87] | -0.26 [-0.94 to 0.42]
Statistical Analysis 1: Comparison: Part 2: Risdiplam vs Part 2: Placebo; Test type: Superiority — The variables included in the MMRM model are: baseline total score, treatment, age group, visit, treatment-by-visit and baseline score-by-visit interaction; p = 0.1328, Mixed Model Repeated Measure Analysis; Least Square Mean Difference = 0.64, 95% CI 2-sided [-0.20 to 1.47]

13. Secondary Outcome: Part 2: Change From Baseline in the MFM-32 Domain 2 (D2) Score at Month 12
Description: The MFM32 comprises 32 items that evaluate physical function in three dimensions: D1 function related to standing and transfer; D2 axial and proximal function; D3 distal motor function. Tasks are scored with a 4-point Likert scale: 0 - cannot initiate the task or maintain the starting position; 1 - performs the task partially; 2 - performs the task incompletely or imperfectly; 3 - performs the task fully and "normally". The D2 items score are summed and expressed on 0-100 scale for the MFM D2 total score. Higher scores indicate increased motor function. A positive change from Baseline indicates improvement. MMRM analysis was performed based on efficacy hypothetical estimand, which included participants data assuming no prohibited medication intended for treatment of SMA was received and participants continued on their randomized treatment until the analysis time point at Month 12.
Time Frame: Baseline (Day-1) and Month 12
Population: The intent-to-treat (ITT) population defined as all randomized participants in Part 2. Participants with missing MFM32 D2 score at Baseline were not included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 118 | 60
Scores on a Scale | 1.04 [-0.38 to 2.46] | -0.93 [-2.87 to 1.02]
Statistical Analysis 1: Comparison: Part 2: Risdiplam vs Part 2: Placebo; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.1030, Mixed Model Repeated Measure Analysis; Least Square Mean Difference = 1.97, 95% CI 2-sided [-0.40 to 4.34]

14. Secondary Outcome: Part 2: Change From Baseline in the MFM-32 Domain 3 (D3) Score at Month 12
Description: The MFM32 comprises 32 items that evaluate physical function in three dimensions: D1 function related to standing and transfer; D2 axial and proximal function; D3 distal motor function. Tasks are scored with a 4-point Likert scale: 0 - cannot initiate the task or maintain the starting position; 1 - performs the task partially; 2 - performs the task incompletely or imperfectly; 3 - performs the task fully and "normally". The D3 items score are summed and expressed on 0-100 scale for the MFM D3 total score. Higher scores indicate increased motor function. A positive change from Baseline indicates improvement. MMRM analysis was performed based on efficacy hypothetical estimand, which included participants data assuming no prohibited medication intended for treatment of SMA was received and participants continued on their randomized treatment until the analysis time point at Month 12.
Time Frame: Baseline (Day-1) and Month 12
Population: The intent-to-treat (ITT) population defined as all randomized participants in Part 2. Participants with missing MFM32 D3 score at Baseline were not included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 115 | 59
Scores on a Scale | 3.68 [2.31 to 5.04] | 1.34 [-0.54 to 3.22]
Statistical Analysis 1: Comparison: Part 2: Risdiplam vs Part 2: Placebo; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.0451, Mixed Model Repeated Measure Analysis; Least Square Mean Difference = 2.34, 95% CI 2-sided [0.05 to 4.62]

15. Secondary Outcome: Part 2: Change From Baseline in the Total Combined Scores of MFM-32 Domains 1 and 2 at Month 12
Description: The MFM32 comprises 32 items that evaluate physical function in three dimensions: D1 function related to standing and transfer; D2 axial and proximal function; D3 distal motor function. Tasks are scored with a 4-point Likert scale: 0 - cannot initiate the task or maintain the starting position; 1 - performs the task partially; 2 - performs the task incompletely or imperfectly; 3 - performs the task fully and "normally". The D1+D2 items score are summed and expressed on 0-100 scale for the MFM D1+D2 total score. Higher scores indicate increased motor function. A positive change from Baseline indicates improvement. MMRM analysis was performed based on efficacy hypothetical estimand, which included participants data assuming no prohibited medication intended for treatment of SMA was received and participants continued on their randomized treatment until the analysis time point at Month 12.
Time Frame: Baseline (Day-1) and Month 12
Population: The intent-to-treat (ITT) population defined as all randomized participants in Part 2. Participants with missing MFM32 D1+D2 scores at Baseline were not included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 118 | 60
Scores on a Scale | 0.69 [-0.07 to 1.45] | -0.59 [-1.64 to 0.45]
Statistical Analysis 1: Comparison: Part 2: Risdiplam vs Part 2: Placebo; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.0489, Mixed Model Repeated Measure Analysis; Least Square Mean Difference = 1.28, 95% CI 2-sided [0.01 to 2.56]

16. Secondary Outcome: Part 2: Change From Baseline in the Total Combined Scores of MFM-32 Domains 2 and 3 at Month 12
Description: The MFM32 comprises 32 items that evaluate physical function in three dimensions: D1 function related to standing and transfer; D2 axial and proximal function; D3 distal motor function. Tasks are scored with a 4-point Likert scale: 0 - cannot initiate the task or maintain the starting position; 1 - performs the task partially; 2 - performs the task incompletely or imperfectly; 3 - performs the task fully and "normally". The D2+D3 items score are summed and expressed on 0-100 scale for the MFM D2+D3 total score. Higher scores indicate increased motor function. A positive change from Baseline indicates improvement. MMRM analysis was performed based on efficacy hypothetical estimand, which included participants data assuming no prohibited medication intended for treatment of SMA was received and participants continued on their randomized treatment until the analysis time point at Month 12.
Time Frame: Baseline (Day-1) and Month 12
Population: The intent-to-treat (ITT) population defined as all randomized participants in Part 2. Participants with missing MFM32 D2+D3 scores at Baseline were not included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 115 | 59
Scores on a Scale | 2.02 [0.84 to 3.20] | -0.14 [-1.76 to 1.48]
Statistical Analysis 1: Comparison: Part 2: Risdiplam vs Part 2: Placebo; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.0326, Mixed Model Repeated Measure Analysis; Least Square Mean Difference = 2.16, 95% CI 2-sided [0.18 to 4.14]

17. Secondary Outcome: Part 2: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) at Month 12 in Participants Aged 6-25 Years
Description: Spirometry is a pulmonary function test that assesses how the lungs work by measuring how much air moves through the airways. Spirometry was performed by all participants aged 6 or older. Forced expiratory volume (FEV1) is the volume forcefully exhaled in the first second of the forced vital capacity test. The best % predicted value out of all attempts were used for the analysis. MMRM analysis was performed based on efficacy hypothetical estimand, which included participants data assuming no prohibited medication intended for treatment of SMA was received and participants continued on their randomized treatment until the analysis time point at Month 12.
Time Frame: Baseline (Day-1) and Month 12
Population: The intent-to-treat (ITT) population defined as all randomized participants in Part 2. Participants with missing FEV1 data at Baseline were not included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Predicted
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 83 | 40
Percentage Predicted | -4.22 [-7.49 to -0.96] | -1.35 [-5.91 to 3.20]
Statistical Analysis 1: Comparison: Part 2: Risdiplam vs Part 2: Placebo; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.3029, Mixed Model Repeated Measure Analysis; Least Square Mean Difference = -2.87, 95% CI 2-sided [-8.36 to 2.62]

18. Secondary Outcome: Part 2: Change From Baseline in the Peak Cough Flow (PCF) at Month 12 in Participants Aged 6-25 Years
Description: Spirometry is a pulmonary function test that assesses how the lungs work by measuring how much air moves through the airways. Spirometry was performed by all participants aged 6 or older. Peak cough flow (PCF) is an assessment of cough strength. The best % predicted value out of all attempts were used for the analysis MMRM analysis was performed based on efficacy hypothetical estimand, which included participants data assuming no prohibited medication intended for treatment of SMA was received and participants continued on their randomized treatment until the analysis time point at Month 12.
Time Frame: Baseline (Day-1) and Month 12
Population: The intent-to-treat (ITT) population defined as all randomized participants in Part 2. Participants with missing PCF data at Baseline were not included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Predicted
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 83 | 42
Percent Predicted | 1.06 [-1.18 to 3.31] | -0.22 [-3.27 to 2.83]
Statistical Analysis 1: Comparison: Part 2: Risdiplam vs Part 2: Placebo; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.4937, Mixed Model Repeated Measure Analysis; Least Square Mean Difference = 1.28, 95% CI 2-sided [-2.42 to 4.99]

19. Secondary Outcome: Part 2: Change From Baseline in the Best Sniff Nasal Inspiratory Pressure (SNIP) at Month 12
Description: The Sniff Nasal Inspiratory Pressure (SNIP) is a volitional, non-invasive test of inspiratory muscle strength that has been successfully applied to children > 2 years of age. Advantages include the simplicity of the maneuver and the absence of a mouthpiece, which is particularly helpful for participants with SMA, who may have bulbar weakness. SNIP also has the advantage of measuring inspiratory pressure during a natural maneuver that is easily performed even by young children with neuromuscular disorders. The best % predicted value out of all attempts were used for the analysis. MMRM analysis was performed based on efficacy hypothetical estimand, which included participants data assuming no prohibited medication intended for treatment of SMA was received and participants continued on their randomized treatment until the analysis time point at Month 12.
Time Frame: Baseline (Day-1) and Month 12
Population: The intent-to-treat (ITT) population defined as all randomized participants in Part 2. Participants with missing SNIP data at Baseline were not included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Predicted
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 118 | 59
Percentage Predicted | 3.42 [0.22 to 6.62] | 1.07 [-3.42 to 5.57]
Statistical Analysis 1: Comparison: Part 2: Risdiplam vs Part 2: Placebo; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.3967, Mixed Model Repeated Measure Analysis; Least Square Mean Difference = 2.35, 95% CI 2-sided [-3.11 to 7.80]

20. Secondary Outcome: Part 2: Change From Baseline in Maximal Inspiratory Pressure (MIP) at Month 12 in Participants Aged 6-25 Years
Description: The maximal inspiratory pressure (MIP) is a non-invasive test of muscle strength, which measures the maximum strength of the diaphragm and other inspiratory muscles. MIP was measured in participants aged 6 or older. Participants were asked to perform a forceful inspiration against an occluded mouth piece. The best % predicted value out of all attempts were used for the analysis. MMRM analysis was performed based on efficacy hypothetical estimand, which included participants data assuming no prohibited medication intended for treatment of SMA was received and participants continued on their randomized treatment until the analysis time point at Month 12.
Time Frame: Baseline (Day-1) and Month 12
Population: The intent-to-treat (ITT) population defined as all randomized participants in Part 2. Participants with missing MIP data at Baseline were not included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Predicted
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 81 | 40
Percentage Predicted | 1.99 [-6.13 to 10.11] | -0.97 [-12.33 to 10.38]
Statistical Analysis 1: Comparison: Part 2: Risdiplam vs Part 2: Placebo; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.6704, Mixed Model Repeated Measure Analysis; Least Square Mean Difference = 2.96, 95% CI 2-sided [-10.78 to 16.70]

21. Secondary Outcome: Part 2: Change From Baseline in Maximal Expiratory Pressure (MEP) at Month 12 in Participants Aged 6-25 Years
Description: The maximal expiratory pressure (MEP) is a non-invasive test of muscle strength, which measures the maximum strength of the abdominal muscles and other expiratory muscles. MEP was measured in participants aged 6 or older. Participants were asked to perform a forceful inspiration against an occluded mouth piece. The best % predicted value out of all attempts were used for the analysis. MMRM analysis was performed based on efficacy hypothetical estimand, which included participants data assuming no prohibited medication intended for treatment of SMA was received and participants continued on their randomized treatment until the analysis time point at Month 12.
Time Frame: Baseline (Day-1) and Month 12
Population: The intent-to-treat (ITT) population defined as all randomized participants in Part 2. Participants with missing MEP data at Baseline were not included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Predicted
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 83 | 41
Percentage Predicted | -2.75 [-6.22 to 0.72] | -2.33 [-7.21 to 2.56]
Statistical Analysis 1: Comparison: Part 2: Risdiplam vs Part 2: Placebo; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.8856, Mixed Model Repeated Measure Analysis; Least Square Mean Difference = -0.43, 95% CI 2-sided [-6.30 to 5.45]

22. Secondary Outcome: Part 2: Change From Baseline in the Participant-Reported SMA Independence Scale (SMAIS) Total Score at Month 12
Description: The SMAIS was developed specifically for SMA participants in order to assess function-related independence. It contains 29 items, assessing the amount of assistance required from another individual to perform daily activities such as eating, or bathing. Each item is scored on a 0-4 scale (with an additional option to indicate that an item is non-applicable). The SMAIS total score ranging from 0-44 is obtained based on 22 items with each item on the 0-2 scale. Lower scores indicate greater dependence on another individual. The SMAIS was completed by participants aged 12 years or older and caregivers of participants aged 2-25 years. MMRM analysis was performed based on efficacy hypothetical estimand, which included participants data assuming no prohibited medication intended for treatment of SMA was received and participants continued on their randomized treatment until the analysis time point at Month 12.
Time Frame: Baseline (Day-1) and Month 12
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 43 | 23
Scores on a Scale | 1.04 [-0.26 to 2.35] | -0.40 [-2.13 to 1.32]
Statistical Analysis 1: Comparison: Part 2: Risdiplam vs Part 2: Placebo; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.1778, Mixed Model Repeated Measure Analysis; Least Square Mean Difference = 1.45, 95% CI 2-sided [-0.68 to 3.57]

23. Secondary Outcome: Part 2: Percentage of Participants Rated by Clinicians as No Change or Improved in the Clinical Global Impression of Change (CGI-C) Scale Ratings at Month 12
Description: The CGI-C is used to score a clinician's impression of a participant's change in global health. It is a single item measure of change in global health, using seven response options: "very much improved", "much improved", "minimally improved", "no change", "minimally worse", "much worse", and "very much worse". Participants considered as "no change or improved" included responses of "no change", "very much improved", "much improved" and "minimally improved". Logistic regression analysis was performed based on efficacy hypothetical estimand, which included participants data assuming no prohibited medication intended for treatment of SMA was received and participants continued on their randomized treatment until the analysis time point at Month 12.
Time Frame: At Month 12
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 120 | 60
Percentage of Participants | 85.8 [79.18 to 92.49] | 83.3 [73.07 to 93.60]
Statistical Analysis 1: Comparison: Part 2: Risdiplam vs Part 2: Placebo; CGI No Change or Improved; Test type: Superiority — [test comment as in outcome 10, analysis 1]; p = 0.6636, Wald-test; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.52 to 2.83]

24. Secondary Outcome: Part 2: Percentage of Participants Who Experience at Least One Disease-Related Adverse Event at Month 12
Description: Disease-related adverse events (AEs) were identified by applying two different types of baskets to the AE dataset: Narrow prospectively defined baskets of MedDRA lowest level terms. This basket was defined based on a group of CDC terms selected from an age and gender matched case control study comparing CDC code rates observed in participants with and without SMA using commercially available insurance claim data (CLAIMS and Market scan data). The lowest level terms included in each basket, coded using the latest version of MedDRA; Broad prospectively defined basket with events selected at preferred term level from all AEs reported in ongoing clinical trials up to January 2019, i.e., prior to unblinding of Part 2 of Study BP39055.
Time Frame: Baseline up to Month 12 (Week 52; up to CCOD of 06 September 2019)
Population: The intent-to-treat (ITT) population defined as all randomized participants in Part 2.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 120 | 60
Percentage of Participants
  Narrow Basket AEs | 46.7 [37.51 to 55.99] | 53.3 [40.00 to 66.33]
  Broad Basket AEs | 65.0 [55.76 to 73.48] | 60.0 [46.54 to 72.44]

25. Secondary Outcome: Part 2: Number of Disease-related Adverse Events Per Patient-years at Month 12
Description: Disease-related AEs were collected through the AE reporting of the study, and the disease-related AE rate was adjusted for patient years (AE rate per 100 patient-years). They were identified by applying two different types of baskets to the AE dataset: Narrow prospectively defined baskets of MedDRA lowest level terms and Broad prospectively defined basket with events selected at preferred term level from all AEs reported in ongoing clinical trials up to January 2019, i.e., prior to unblinding of Part 2 of Study BP39055.
Time Frame: Baseline up to Month 12 (Week 52; up to CCOD of 06 September 2019)
Population: The intent-to-treat (ITT) population defined as all randomized participants in Part 2.
Measure: Number (95% Confidence Interval); unit: Number of Events per 100 Patient-Years
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 120 | 60
Number of Events per 100 Patient-Years
  Narrow Basket AEs | 101.51 [84.23 to 121.29] | 119.77 [93.71 to 150.82]
  Broad Basket AEs | 217.29 [191.63 to 245.42] | 199.61 [165.50 to 238.68]

26. Secondary Outcome: Part 2: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) in the Placebo-Controlled Period
Description: An adverse event (AE) is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Day 1 up to 12 months of the placebo-controlled period
Population: All participants in Part 2 who receive at least one dose of study medication (risdiplam or placebo) were included in the safety population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 120 | 60
Percentage of Participants
  With at Least One AE | 92.5 | 91.7
  With at Least One SAE | 20.0 | 18.3

27. Secondary Outcome: Part 2: Percentage of Participants With Treatment Discontinuation Due to Adverse Events (AEs) and Serious Adverse Events (SAEs) in the Placebo-Controlled Period
Description: as for outcome 26
Time Frame: Day 1 up to 12 months of the placebo-controlled period
Population: All participants in Part 2 who received at least one dose of study medication (risdiplam or placebo) were included in the safety population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 120 | 60
Percentage of Participants
  Due to AE | 0.0 | 0.0
  Due to SAE | 0.0 | 0.0

28. Secondary Outcome: Part 2: Number of Participants Aged 6-25 Years With Suicidal Ideation Based on Columbia-Suicide Severity Rating Scale (C-SSRS) in the Placebo-Controlled Period
Description: The Columbia Suicide Severity Rating Scale (C-SSRS) is used to assess the lifetime suicidality of a participant (C-SSRS baseline) as well as any new instances of suicidality (C-SSRS since last visit). The structured interview prompts recollection of suicidal ideation, including the intensity of the ideation, behavior, and attempts with actual/potential lethality. The C-SSRS assessments results were collected for participants aged 6 years and older.
Time Frame: Day 1 up to 12 months of the placebo-controlled period
Population: The intent-to-treat (ITT) population defined as all randomized participants in Part 2. Data was collected for participants aged 6-25 years.
Measure: Number; unit: Number of Participants
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 83 | 42
Number of Participants
  Wish to be Dead | 1 | 1
  Non-specific Active Suicidal Thoughts | 1 | 1
  Ideation with Any Methods, No Intent to Act | 1 | 1
  Ideation with Some Intent to Act, No Plan | 0 | 1
  Ideation with Specific Plan and Intent | 0 | 1

29. Secondary Outcome: Part 2: Number of Participants Aged 6-25 Years With Suicidal Behavior Based on Columbia-Suicide Severity Rating Scale (C-SSRS) in the Placebo-Controlled Period
Description: as for outcome 28
Time Frame: Day 1 up to 12 months of the placebo-controlled period
Population: as for outcome 28
Measure: Number; unit: Number of Participants
Arm/Group | Part 2: Risdiplam | Part 2: Placebo
Number analyzed (Participants) | 83 | 42
Number of Participants
  Preparatory Acts or Behavior | 0 | 0
  Aborted Attempt | 0 | 0
  Interrupted Attempt | 0 | 0
  Actual Attempt (non-fatal) | 0 | 0
  Completed Suicide | 0 | 0

30. Secondary Outcome: Median Fold Change From Baseline in Survival of Motor Neuron (SMN) Protein Levels in Blood
Time Frame: Part 1: Day -1, pre-dose of Weeks 1, 2 (>/= 12 years only), 17, 35 and 104, and at 4h post-dose of Weeks 4 and 52. Part 2: Day -1, pre-dose of Weeks 1, 17, 35 and 104, and at 4h post-dose of Weeks 4 and 52.
Population: All participants with at least one time point with a protein measurement were included in the pharmacodynamic (PD) analysis data set.
Measure: Median (Full Range); unit: unitless
Groups:
- Part 2: All Risdiplam: Children aged 2-11 years and adolescent and adult participants aged 12-25 years received risdiplam or risdiplam matching placebo.
Arm/Group | Part 1: All Risdiplam | Part 2: All Risdiplam
Number analyzed (Participants) | 51 | 169
unitless | 2.91 [2.14 to 4.18] | 1.96 [0.2 to 4.48]

31. Secondary Outcome: Part 1 and 2: Maximum Plasma Concentration (Cmax) of Risdiplam at Year 5
Description: Reported here is the maximum observed concentration throughout the observation period.
Time Frame: Day 1: 1, 2, 4, 6 h postdose, Weeks 4, 8 (Part 1 only), 52, 87: pre-dose, 1, 2, 4, 6 h post-dose and Weeks 1 (Day 7), 2, 8 (Part 2 only) 17, 35, 70, 104: predose
Population: All participants with at least one time point with a risdiplam concentration measurement were included in the pharmacokinetic (PK) analysis data set.
Measure: Median (Full Range); unit: nanograms/milliliter (ng/mL)
Arm/Group | Part 1: All Risdiplam | Part 2: All Risdiplam
Number analyzed (Participants) | 51 | 179
nanograms/milliliter (ng/mL) | 137 [58.2 to 242] | 140 [42.7 to 313]

32. Secondary Outcome: Part 1 and 2: Area Under the Curve (AUC) From 0 to 24 Hours of Risdiplam at Year 5 Visit
Time Frame: Year 5 visit pre-dose, 1, 2, 4, 6, 24 hours post-dose
Population: All participants with at least one time point with a risdiplam concentration measurement were included in the PK analysis data set.
Measure: Median (Full Range); unit: ng*h/mL
Arm/Group | Part 1: All Risdiplam | Part 2: All Risdiplam
Number analyzed (Participants) | 49 | 160
ng*h/mL | 1700 [1160 to 2590] | 1880 [1200 to 2890]

33. Secondary Outcome: Part 1 and 2: Concentration at the End of a Dosing Interval (Ctrough) of Risdiplam at Year 5
Time Frame: The last predose sample collected from each participant who had at least 1400 days of risdiplam treatment duration.
Population: as for outcome 32
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Part 1: All Risdiplam | Part 2: All Risdiplam
Number analyzed (Participants) | 49 | 107
ng/mL | 54.1 [21.3 to 108] | 57.2 [4.50 to 229]

ADVERSE EVENTS:
Time Frame: Part 1 and Part 2: Up to approximately 5 years
Description: The safety population included all participants who received at least one dose of study medication (risdiplam or placebo) whether prematurely withdrawn or not.
Groups:
- Part 1 Group A: Adolescents and Adults (3 mg Risdiplam); Part 1 Group A: Adolescents and Adults (5 mg Risdiplam): Adolescent and adult participants aged 12-25 years received risdiplam for at least 12 weeks during the placebo-controlled period.
- Part 1 Group A: Adolescents and Adults (Placebo-Control Period Pooled): Adolescent and adult participants aged 12-25 years received placebo matching to risdiplam for at least 12 weeks during the placebo-controlled period.
- Part 1 Group B: Children (0.02 mg/kg Risdiplam); Part 1 Group B: Children (0.05 mg/kg Risdiplam); Part 1 Group B: Children (0.15 mg/kg Risdiplam); Part 1 Group B: Children (0.25 mg/kg Risdiplam): Children aged 2-11 years received risdiplam for at least 12 weeks during the placebo-controlled period.
- Part 1 Group B: Children (Placebo-Control Period Pooled): Children aged 2-11 years received placebo matching to risdiplam for at least 12 weeks during the placebo-controlled period.
- Part 2 Placebo-Controlled: Risdiplam: Participants aged 2-25 years received risdiplam at the dose of 5 mg once daily for participants with a body weight (BW) >/=20kg or 0.25 mg/kg for participants with a BW <20 kg for 12 months during the placebo-controlled period..
- Part 2 Placebo-Controlled: Placebo: Participants aged 2-25 years received placebo matching to risdiplam for 12 months during the placebo-controlled period.
- Part 2 OLT: Risdiplam/Risdiplam: Once the Part 2 placebo-controlled period was completed participants received risdiplam at the dose of 5 mg once daily for participants with a body weight (BW) >/=20kg or 0.25 mg/kg for participants with a BW <20 kg for another 12 months (Month 12-24) in the open-label treatment (OLT) phase.
- Part 2 OLT: Placebo/Risdiplam: Once the Part 2 placebo-controlled period was completed participants switched to risdiplam at the dose of 5 mg once daily for participants with a body weight (BW) >/=20kg or 0.25 mg/kg for participants with a BW <20 kg for 12 months (Month 12-24) in the open-label treatment (OLT) phase.
- Part 2 OLE: Risdiplam: Once the Part 2 OLT period ended participants entered the open-label extension period and continued to receive risdiplam at the dose of 5 mg once daily for participants with a body weight (BW) >/=20kg or 0.25 mg/kg for participants with a BW <20 kg.
Arm/Group | Part 1 Group A: Adolescents and Adults (3 mg Risdiplam) | Part 1 Group A: Adolescents and Adults (5 mg Risdiplam) | Part 1 Group A: Adolescents and Adults (Placebo-Control Period Pooled) | Part 1 Group B: Children (0.02 mg/kg Risdiplam) | Part 1 Group B: Children (0.05 mg/kg Risdiplam) | Part 1 Group B: Children (0.15 mg/kg Risdiplam) | Part 1 Group B: Children (0.25 mg/kg Risdiplam) | Part 1 Group B: Children (Placebo-Control Period Pooled) | Part 1 Group A: OLE | Part 1 Group B: OLE | Part 2 Placebo-Controlled: Risdiplam | Part 2 Placebo-Controlled: Placebo | Part 2 OLT: Risdiplam/Risdiplam | Part 2 OLT: Placebo/Risdiplam | Part 2 OLE: Risdiplam
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/6 | 0/7 | 0/14 | 0/21 | 0/7 | 0/10 | 0/20 | 0/31 | 0/120 | 0/60 | 0/117 | 0/59 | 1/175
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10 | 0/6 | 0/7 | 0/14 | 0/21 | 0/7 | 1/10 | 5/20 | 9/31 | 24/120 | 11/60 | 25/117 | 4/59 | 34/175
Other Adverse Events (participants affected / at risk) | 9/10 | 8/10 | 4/6 | 6/7 | 12/14 | 18/21 | 6/7 | 9/10 | 17/20 | 28/31 | 101/120 | 50/60 | 88/117 | 40/59 | 140/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Group A: Adolescents and Adults (3 mg Risdiplam) (N=10) | Part 1 Group A: Adolescents and Adults (5 mg Risdiplam) (N=10) | Part 1 Group A: Adolescents and Adults (Placebo-Control Period Pooled) (N=6) | Part 1 Group B: Children (0.02 mg/kg Risdiplam) (N=7) | Part 1 Group B: Children (0.05 mg/kg Risdiplam) (N=14) | Part 1 Group B: Children (0.15 mg/kg Risdiplam) (N=21) | Part 1 Group B: Children (0.25 mg/kg Risdiplam) (N=7) | Part 1 Group B: Children (Placebo-Control Period Pooled) (N=10) | Part 1 Group A: OLE (N=20) | Part 1 Group B: OLE (N=31) | Part 2 Placebo-Controlled: Risdiplam (N=120) | Part 2 Placebo-Controlled: Placebo (N=60) | Part 2 OLT: Risdiplam/Risdiplam (N=117) | Part 2 OLT: Placebo/Risdiplam (N=59) | Part 2 OLE: Risdiplam (N=175)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (4)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 2 (4)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 10 (12) | 2 (2) | 8 (10) | 0 (0) | 8 (12)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Near drowning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cryptorchism (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malpositioned teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ill-defined disorder (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infective thrombosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lymph gland infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Febrile convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device breakage (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Encopresis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part 1 Group A: Adolescents and Adults (3 mg Risdiplam) (N=10) | Part 1 Group A: Adolescents and Adults (5 mg Risdiplam) (N=10) | Part 1 Group A: Adolescents and Adults (Placebo-Control Period Pooled) (N=6) | Part 1 Group B: Children (0.02 mg/kg Risdiplam) (N=7) | Part 1 Group B: Children (0.05 mg/kg Risdiplam) (N=14) | Part 1 Group B: Children (0.15 mg/kg Risdiplam) (N=21) | Part 1 Group B: Children (0.25 mg/kg Risdiplam) (N=7) | Part 1 Group B: Children (Placebo-Control Period Pooled) (N=10) | Part 1 Group A: OLE (N=20) | Part 1 Group B: OLE (N=31) | Part 2 Placebo-Controlled: Risdiplam (N=120) | Part 2 Placebo-Controlled: Placebo (N=60) | Part 2 OLT: Risdiplam/Risdiplam (N=117) | Part 2 OLT: Placebo/Risdiplam (N=59) | Part 2 OLE: Risdiplam (N=175)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0/0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 3 (4) | 2 (2) | 5 (5) | 2 (2) | 3 (4)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal infiltrates (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema eyelids (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Retinal dystrophy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (1) | 2 (2) | 4 (6) | 8 (10) | 5 (6) | 7 (10) | 4 (5) | 7 (15)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 3 (5) | 7 (7) | 2 (3) | 1 (1) | 1 (1) | 9 (10)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (12) | 9 (10) | 3 (3) | 4 (4) | 2 (4) | 8 (9)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (14) | 21 (27) | 5 (5) | 10 (12) | 6 (8) | 17 (26)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip pruritus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (3) | 3 (4) | 11 (13) | 3 (4) | 4 (5) | 3 (6) | 8 (10)
Oral mucosal erythema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue oedema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 4 (6) | 5 (7) | 1 (1) | 1 (1) | 4 (6) | 10 (27) | 17 (35) | 14 (22) | 15 (31) | 9 (13) | 20 (43)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Granuloma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperpyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 6 (6)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 2 (4) | 1 (2) | 0 (0) | 2 (2) | 3 (4) | 4 (5) | 1 (1) | 3 (5) | 9 (19) | 18 (52) | 25 (41) | 10 (20) | 15 (22) | 6 (7) | 30 (38)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 7 (15) | 7 (9) | 10 (12) | 6 (7) | 4 (4) | 9 (11)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 9 (12) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 55 (60)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (6) | 3 (3) | 1 (1) | 2 (3) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 3 (5) | 0 (0) | 1 (2) | 1 (1) | 1 (3)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 3 (3)
Ear infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (1) | 4 (7) | 9 (11) | 7 (10) | 5 (6) | 9 (9) | 5 (7) | 12 (18)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 3 (5)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Groin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (12) | 6 (8) | 3 (3) | 3 (4) | 3 (3) | 2 (2) | 8 (8)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Laryngitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 3 (7) | 12 (23) | 31 (54) | 15 (21) | 26 (34) | 6 (7) | 34 (48)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (3) | 4 (4) | 6 (8) | 3 (3) | 6 (6) | 4 (4) | 7 (7)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 5 (6) | 3 (3) | 2 (2) | 0 (0) | 12 (16)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 8 (10) | 6 (9) | 7 (8) | 1 (1) | 5 (5)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 5 (10) | 3 (4) | 1 (1) | 3 (3) | 7 (7)
Scarlet fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (4) | 2 (4) | 1 (1) | 2 (2) | 5 (10)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (5) | 2 (3) | 0 (0) | 3 (10) | 14 (47) | 38 (54) | 18 (27) | 18 (24) | 10 (18) | 49 (99)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (7) | 6 (7) | 0 (0) | 2 (3) | 2 (2) | 12 (21)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 2 (4) | 2 (2) | 5 (6) | 5 (5)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 3 (3)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (2) | 2 (2) | 1 (1) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Tooth dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric pH decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 5 (6) | 6 (9) | 0 (0) | 3 (3) | 2 (2) | 13 (21)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (14) | 2 (3) | 3 (4) | 2 (4) | 3 (3) | 1 (1) | 11 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (13) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 4 (4) | 1 (3) | 2 (2) | 3 (3) | 10 (12)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 7 (7)
Headache (Nervous system disorders) | 1 (3) | 1 (3) | 0 (0) | 1 (18) | 1 (18) | 2 (20) | 1 (2) | 0 (0) | 3 (60) | 6 (47) | 24 (88) | 10 (23) | 12 (76) | 11 (32) | 20 (84)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Initial insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 2 (7) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (27) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Premenstrual pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (4) | 1 (2) | 2 (4) | 4 (5) | 11 (31) | 17 (27) | 12 (19) | 12 (16) | 5 (7) | 14 (19)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4) | 1 (1) | 1 (2) | 1 (2) | 1 (2) | 0 (0) | 1 (2) | 3 (6) | 6 (8) | 6 (6) | 7 (8) | 4 (4) | 1 (1) | 11 (16)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (7) | 6 (6) | 3 (3) | 3 (4) | 1 (1) | 10 (12)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (5) | 4 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (4) | 3 (5) | 1 (1) | 3 (4) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 5 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (5)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 5 (5) | 1 (1) | 3 (3) | 1 (1) | 5 (6)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 9 (11) | 1 (1) | 6 (6) | 0 (0) | 7 (10)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT02908685/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT02908685/SAP_002.pdf